CLINICAL TRIAL: NCT00052091
Title: PST in Geriatric Depression With Executive Dysfunction
Brief Title: Therapy for Depressed Elders With Thought Problems
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Pat Arean, Professor, Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H7472-19384-8; R01MH063982 (NIH); DATR A4-GPS
Record Dates: First submitted 2003-01-22; First posted 2003-01-23 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Depression; Cognition Disorders
Keywords: Geriatrics
MeSH Terms: conditions — Depression; Cognition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Problem Solving Therapy (Experimental): 12 weekly sessions of problem solving therapy (PST)
  Interventions: Behavioral: Problem Solving Therapy
- 2 Brief Supportive Therapy (Experimental): 12 weekly sessions of brief supportive therapy (BST)
  Interventions: Behavioral: Brief Supportive Therapy

INTERVENTIONS:
Behavioral: Problem Solving Therapy — A 12 week cognitive behavioral intervention for depression that teaches patients a structured approach to solving social problems.
  Arms: 1 Problem Solving Therapy
Behavioral: Brief Supportive Therapy — A 12 week intervention for depression that focuses on supporting patients attempts to cope with depression.
  Arms: 2 Brief Supportive Therapy

SUMMARY:
This study will compare the effectiveness of Problem Solving Therapy and Brief Supportive Therapy in treating elderly patients with major depression and thought problems.

DETAILED DESCRIPTION:
Patients who suffer from a combination of major depression and executive dysfunction symptoms often respond poorly to treatment with antidepressants. It is important, therefore, to find effective alternative therapies to treat these symptoms.

Patients are randomly assigned to receive 12 sessions (1 session/week for 12 weeks) of either PST or BST. Following treatment, patients are followed for 6 months to determine functional and clinical outcomes. Depression scales, disability scales, and scales that measure problem solving skills are used to assess patients.

ELIGIBILITY:
Inclusion Criteria:

* Nonpsychotic, unipolar major depression
* Cognitive impairment
* English speaking

Exclusion Criteria:

* High suicide risk
* Dementia
* Acute or severe medical illness
* Current psychotherapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2002-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression | Measured at screening, weeks 1 through 12, and week 36

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A. Arean, PhD, Principal Investigator — University of California at San Francisco
Locations (2):
- United States (2):
  - University of California at San Francisco, San Francisco, California
  - Weill Medical College of Cornell University, White Plains, New York

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Arean PA, Raue P, Mackin RS, Kanellopoulos D, McCulloch C, Alexopoulos GS. Problem-solving therapy and supportive therapy in older adults with major depression and executive dysfunction. Am J Psychiatry. 2010 Nov;167(11):1391-8. doi: 10.1176/appi.ajp.2010.09091327. Epub 2010 Jun 1. PMID 20516155
- [Result] Alexopoulos GS, Raue PJ, Kiosses DN, Mackin RS, Kanellopoulos D, McCulloch C, Arean PA. Problem-solving therapy and supportive therapy in older adults with major depression and executive dysfunction: effect on disability. Arch Gen Psychiatry. 2011 Jan;68(1):33-41. doi: 10.1001/archgenpsychiatry.2010.177. PMID 21199963
- [Derived] Solomonov N, Kerchner D, Bein O, Lee CE, Diaz JL, Ciarleglio A, Kim S, Sirey JA, Gunning FM, Raue PJ, Banerjee S, Arean PA, Alexopoulos GS. Precision Assignment to Psychosocial Interventions for Late-Life Depression: An Automated Treatment Decision Rule. JAMA Psychiatry. 2025 Nov 1;82(11):1075-1084. doi: 10.1001/jamapsychiatry.2025.2518. PMID 40960814
- [Derived] Alexopoulos GS, O'Neil R, Banerjee S, Raue PJ, Victoria LW, Bress JN, Pollari C, Arean PA. "Engage" therapy: Prediction of change of late-life major depression. J Affect Disord. 2017 Oct 15;221:192-197. doi: 10.1016/j.jad.2017.06.037. Epub 2017 Jun 19. PMID 28647669
- [Derived] Gustavson KA, Alexopoulos GS, Niu GC, McCulloch C, Meade T, Arean PA. Problem-Solving Therapy Reduces Suicidal Ideation In Depressed Older Adults with Executive Dysfunction. Am J Geriatr Psychiatry. 2016 Jan;24(1):11-17. doi: 10.1016/j.jagp.2015.07.010. Epub 2015 Jul 30. PMID 26743100
- [Derived] Alexopoulos GS, Raue PJ, Kiosses DN, Seirup JK, Banerjee S, Arean PA. Comparing engage with PST in late-life major depression: a preliminary report. Am J Geriatr Psychiatry. 2015 May;23(5):506-13. doi: 10.1016/j.jagp.2014.06.008. Epub 2014 Jun 26. PMID 25081818